CLINICAL TRIAL: NCT02468661
Title: A Phase Ib/II, Open-label, Multicenter Trial With Oral cMET Inhibitor INC280 Alone and in Combination With Erlotinib Versus Platinum With Pemetrexed in Adult Patients With EGFR Mutated, cMET-amplified, Locally Advanced/Metastatic Non-small Cell Lung Cancer (NSCLC) With Acquired Resistance to Prior EGFR Tyrosine Kinase Inhibitor (EGFR TKI)
Brief Title: A Safety and Efficacy Study of INC280 Alone, and in Combination With Erlotinib, Compared to Chemotherapy, in Advanced/Metastatic Non-small Cell Lung Cancer Patients With EGFR Mutation and cMET Amplification
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Major challenge for enrollment of participants.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINC280B2201; 2015-001241-84 (EudraCT Number)
Record Dates: First submitted 2015-06-01; First posted 2015-06-11 (Estimated); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; NSCLC; INC280; erlotinib; advanced/metastatic non-small cell lung cancer; EGFR mutation; cMET amplification; EGFR tyrosine kinase inhibitor (EGFR TKI)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Intervention Model Description: The study started as a single assignment study which was to move to a parallel design (3 arms) but the study was stopped after cohort #3 in the phase I part and so never moved into phase 2.
Masking Description: The study started as a non-randomized study, and was to move into randomized part in phase II. However the study was stopped after cohort #3 in the phase I part and so never moved into phase II.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- INC280 200mg BID + ERL 150mg QD (Experimental): Subjects who took INC280 200mg twice a day (BID) in combination with erlotinib (ERL) 150mg one a day (QD)
  Interventions: Drug: INC280 single agent; Drug: erlotinib
- INC280 400mg BID + ERL 150mg QD (Experimental): Subjects who took INC280 400mg twice a day (BID) in combination with erlotinib (ERL) 150mg one a day (QD)
  Interventions: Drug: INC280 single agent; Drug: erlotinib

INTERVENTIONS:
Drug: INC280 single agent
Drug: erlotinib

SUMMARY:
The purpose of this study was to determine the maximum tolerated dose (MTD) or recommended phase II dose (RP2D) of INC280 in combination with erlotinib in the Phase Ib of this study, and to assess the anti-tumor activity and safety of INC280 alone, and in combination with erlotinib, versus platinum with pemetrexed in the Phase II of this study, in adult patients with EGFR mutated, cMET amplified, advanced/metastatic non-small cell lung cancer with acquired resistance to prior EGFR TKI.

DETAILED DESCRIPTION:
The decision was taken to halt study enrollment with Cohort #3 in Phase Ib. Therefore, activities for the planned Phase II were not initiated.

This decision to stop further development of this combination was taken due to the challenge for enrollment in this very rare patient population along with the rapidly evolving disease landscape setting.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic NSCLC
* EGFR mutation (L858R and /or ex19del)
* cMET amplification by FISH (GCN ≥ 6),
* Acquired resistance to EGFR TKI (1st or 2nd generation)
* ECOG performance status (PS) ≤ 1.

Exclusion Criteria:

* Prior treatment with 3rd generation TKI
* PhaseII : Prior treatment with any of the following agents:

  * Crizotinib, or any other cMET inhibitor or HGF-targeting inhibitor.
  * Concomitant EGFR TKI and platinum based chemotherapy as first line regimen.
  * Platinum-based chemotherapy as first line treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Phase Ib: Frequency and characteristics of Dose Limiting Toxicity (DLTs) to the INC280 and erlotinib combination | First 28 days of dosing
  To determine MTD and/or RP2D of INC280 in combination with erlotinib

SECONDARY OUTCOMES:
Phase Ib: Overall response rate (ORR) | Every 3 weeks, up to 5 years
  ORR, proportion of patients with a best overall response of complete response or partial Response (CR+PR)
Phase Ib: Disease Control Rate (DCR) | Every 6 weeks, up to 2 years
  DCR, proportion of patients with best overall response of CR, PR or SD
Phase Ib: Duration of Response (DOR) | Every 6 weeks, up to 2 years
  DOR, defined as time from the first documented CR or PR to first documented progression or death due to any cause
Phase Ib: Progression-free Survival (PFS) | Every 6 weeks, up to 2 years
  PFS, defined as time from the first dose of study treatment to disease progression or death due to any cause
Phase Ib: Number of patients with adverse events (AEs) as a measure of safety and tolerability | Every 3 weeks, up to 2 years
  Safety and tolerability of INC280 in combination with erlotinib assessed by change in vital signs, laboratory results and electrocardiogram (ECG).
Phase Ib: Plasma concentration-time profiles of INC280 and pharmacokinetic parameters | 6 weeks
  Composite pharmacokinetics of INC280 in the presence of erlotinib.
Phase Ib: Plasma concentration-time profiles of erlotinib in the presence of INC280 | 6 weeks
  Composite pharmacokinetics of erlotinib in the presence of INC280.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (32):
- United States (5):
  - Los Angeles Hematology/Oncology Medical Group, Los Angeles, California
  - University of California Irvine Medical Center Chao Family SC, Orange, California
  - Henry Ford Hospital SC, Detroit, Michigan
  - Dartmouth Hitchcock Medical Center SC, Lebanon, New Hampshire
  - Seattle Cancer Care Alliance, Seattle, Washington
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
- France (5):
  - Novartis Investigative Site, Nice, Alpes Maritimes
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Strasbourg
- Germany (3):
  - Novartis Investigative Site, Tübingen, Baden-Wurttemberg
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Berlin
- Italy (6):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Meldola, FC
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Verona, VR
- Japan (4):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Akashi, Hyōgo
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Okayama, Okayama-ken
- NKI-AVL, Department of Thoracic-Oncology, Amsterdam, Netherlands
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (3):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: No